CLINICAL TRIAL: NCT03169413
Title: Human Leucocytic Antigen Typing and Mutation of Adenosine Triphosphate Sensitive Potassium Channel Gene in Diabetic Patients Diagnosed Under the Age of One Year.
Brief Title: Gene Study for Infantile Onset Diabetes
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Shimaa Kamal, Principle Investigator, Assiut University
Other Study IDs: IDM
Record Dates: First submitted 2017-05-25; First posted 2017-05-30 (Actual); Last update posted 2017-05-31 (Actual); Status verified 2017-05

CONDITIONS: Study Genetic Basis of Infantile Onset Diabetes Mellitus

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- cases: Fifty diabetic children diagnosed under the age of one year subjected to genetic analysis to study human leucocytic antigen haplotype class two (DR-DQ) and detection of mutations in the potassium channel, inwardly rectifying subfamily J member 11 gene encoding the Kir6.2 subunit of adenosine triphosphate sensitive potassium channel also possible risk factors associated with the disease.
  Interventions: Genetic: Human Leucocytic antigen typing and mutation of adenosine triphosphate sensitive K channel gene in diabetic patients diagnosed under the age of one year.
- control one: Twenty five diabetic children diagnosed after the age of one year subjected to genetic study to study human leucocytic antigen and possible of presence of gene mutation of the potassium channel, inwardly rectifying subfamily J member 11 gene encoding the Kir6.2 subunit of adenosine triphosphate sensitive potassium channel and possible risk factors associated with disease .
  Interventions: Genetic: Human Leucocytic antigen typing and mutation of adenosine triphosphate sensitive K channel gene in diabetic patients diagnosed under the age of one year.
- control two: Twenty five healthy children matched by age subjected to genetic study to study human leucocytic antigen and possible of presence of gene mutation of the potassium channel, inwardly rectifying subfamily J member 11 gene encoding the Kir6.2 subunit of adenosine triphosphate sensitive potassium channel and exposure to similar risk factors associated with disease .
  Interventions: Genetic: Human Leucocytic antigen typing and mutation of adenosine triphosphate sensitive K channel gene in diabetic patients diagnosed under the age of one year.

INTERVENTIONS:
Genetic: Human Leucocytic antigen typing and mutation of adenosine triphosphate sensitive K channel gene in diabetic patients diagnosed under the age of one year. — Gene study

SUMMARY:
Diabetes mellitus is a group of metabolic diseases characterized by chronic hyperglycemia resulting from defects in insulin secretion, insulin action, or both.

According to American Diabetes Association diabetes can be classified into the following general categories: Type one diabetes (due to beta cell destruction, usually leading to absolute insulin deficiency), Type two diabetes (due to a progressive insulin secretory defect on the background of insulin resistance), Gestational diabetes mellitus and specific types of diabetes due to other causes, example monogenic diabetes syndromes (such as neonatal diabetes and maturity-onset diabetes of the young, diseases of the exocrine pancreas, and drug induced diabetes.

DETAILED DESCRIPTION:
Type one diabetes mellitus is one of the most common endocrine and metabolic conditions in childhood, it accounts for 5-10 percent of all diabetes cases.

Three-quarters of all cases of type one diabetes are diagnosed in individuals under eighteen years of age.

Data on incidence of childhood onset type one diabetes mellitus are very limited. Data from large epidemiological studies worldwide indicate that on an annual basis, the overall increase in the incidence of type one diabetes mellitus is around three percent.

The incidence rate increases from birth and peaks between the ages of ten to fourteen years. There is increase in incidence of type one diabetes mellitus throughout the world is especially, marked in young children, Registries in Europe suggest that incidence of type one diabetes mellitus were highest in the youngest age-group less than four years There is a seasonal pattern in the onset of type one diabetes mellitus with increased cases during late autumn, winter, and early spring.

Although most common autoimmune diseases usually affect females, but girls and boys are equally affected with type one diabetes mellitus in young populations.

The underlying pathophysiological mechanism of the disease is cellular-mediated autoimmune destruction of the pancreatic beta cells, the rate of beta cell destruction is quite variable, being rapid in some individuals (mainly infants and children) and slow in others (mainly adult).

The triggers for the autoimmune attack are not fully understood, but it is now widely accepted that both environmental and genetic factors contribute to it.

The genetic basic of the disease can be explained as the disease involves many genes, the risk of a child developing type one diabetes is about five percent if the father has it, about eight percent if a sibling has it, about three percent if the mother has type one diabetes.

If one identical twin is affected there is about a fifty percent chance the other will also be affected.

Some studies of heritability has estimated it at eighty to eighty sex percent. Depending on locus or combination of loci, they can be dominant, recessive, or somewhere in between. The strongest gene is located in the major histocompatability class two region on chromosome sex, at staining region 6p21. It has been reported that only ten percent of those who are genetically predisposed to type one diabetes mellitus actually develop the disease; however, that percentage appears to be changing and environmental factors may play an increasingly important role in determining risk.

Finally, migration studies show an increased type one diabetes mellitus incidence in population groups who move from an area of low incidence to one of high incidence.

The Possible maternal risk factors for type one diabetes mellitus include maternal age older than twenty five years, cesarean section, high level of education, infants of mothers with body mass index of thirty or higher. or higher, infants of white mothers, and maternal diabetes.

Some studies have reported associations between birth weight and risk of type one diabetes mellitus, being born large for gestational age, and rapid postnatal growth associated with an increased risk for type one diabetes.

Other risk factors include: lack of breast feeding, early introduction of cow milk, and early introduction of gluten containing food before age of four month or late introduction after the age of seven months, lack of vitamin D supplementation during first year of life consumption of sugary foods, exposure to certain viruses as cytomegalovirus, measles, or mumps, childhood vaccination, and maternal-childhood blood group incompatibility.

Neonatal diabetes is a rare cause of hyperglycemia, with an estimated incidence of 1 in 500,000 births.

Two main subgroups are recognized in about equal proportions: permanent neonatal diabetes and transient neonatal diabetes.The latter remits in infancy or early childhood but may recur later in life.

Patients with permanent neonatal diabetes typically have reduced birth weight, a reflection of reduced insulin production in utero, and whilst most are diagnosed with diabetes before sex months a few rare cases have been reported with diabetes diagnosed between sex and twelve months of life. In contrast to Type one diabetes permanent diabetes mellitus is not associated with high risk human leucocytic antigen haplotypes or the presence of pancreatic autoantibodies, and is most commonly due to activating mutations in either of the genes encoding the two subunits of the adenosine triphosphate sensitive potassium channel (potassium channel, inwardly rectifying subfamily J member 11) these mutations also occur in transient neonatal diabetes. In most of these patients, switching from insulin to oral sulfonylurea therapy leads to improved metabolic control.

The diabetes presenting within the first sex months of life is unlikely to represent type one diabetes and usually due to gene mutation, so molecular genetic analysis of this group of patients should be done. Additionally, individuals with a diagnosis of diabetes after sex months-of-age should also receive genetic analysis if their diabetes presentation is atypical for type one diabetes, has features consistent with a known monogenic cause, or if there are additional affected family members with a history of neonatal diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Diabetic patients with disease onset under the age of one year according to American Diabetes Association criteria 2016 which include:
* Fasting plasma glucose level at or above 7 millimol/Litre.
* Plasma glucose at or above 11.1 millimol/Litre two hours after a 1.75 gram/kilogram oral glucose load as in a glucose tolerance test.
* Symptoms of hyperglycemia and random plasma glucose at or above 11.1 millimol/Litre.
* Glycated hemoglobin at or above 48 millimol/mol.

Exclusion Criteria:

-Diabetic children with the disease onset above the age of one year.

Ages: 1 Year to 3 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Diabetic patient diagnosed under the age of one year within two years, 50 randomly chosen patients will subjected to genetic analysis and two control group one will include 25 diabetic patient diagnosed after the age of one year matched by gender and by age (within a few days of birth), the other group include 25 healthy children from the community matched by gender and by age (within a few days of birth).
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2018-01 (Estimated); Primary Completion 2020-01 (Estimated); Study Completion 2020-08 (Estimated)

PRIMARY OUTCOMES:
Human Leucocytic antigen typing and mutation of adenosine triphosphate sensitive potassium channel gene in diabetic patients diagnosed under the age of one year. | At time of diagnosis with diabetes under the age of one year
  Polymerase chain reaction / Deoxyribonucleic acid sequencing

SECONDARY OUTCOMES:
Rate of diabetes mellitus in patients under age of one year attending pediatric endocrinology unit in Pediatric assiut University Hospital | Within two years
  Total coverage of all diabetic cases diagnosed under the age of one year
dentification of possible demographic and environmental risk factors associated with increased risk of diabetes in diabetic patient under the age of one year. | Within two years
  Identification of prenatal, perinatal, natal history,nutritional history, vaccination history and hygiene measures

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Aguilar-Bryan L, Bryan J. Neonatal diabetes mellitus. Endocr Rev. 2008 May;29(3):265-91. doi: 10.1210/er.2007-0029. Epub 2008 Apr 24. PMID 18436707
- [Background] Babenko AP, Polak M, Cave H, Busiah K, Czernichow P, Scharfmann R, Bryan J, Aguilar-Bryan L, Vaxillaire M, Froguel P. Activating mutations in the ABCC8 gene in neonatal diabetes mellitus. N Engl J Med. 2006 Aug 3;355(5):456-66. doi: 10.1056/NEJMoa055068. PMID 16885549
- [Background] Bluestone JA, Herold K, Eisenbarth G. Genetics, pathogenesis and clinical interventions in type 1 diabetes. Nature. 2010 Apr 29;464(7293):1293-300. doi: 10.1038/nature08933. PMID 20432533
- [Background] Noble JA, Valdes AM. Genetics of the HLA region in the prediction of type 1 diabetes. Curr Diab Rep. 2011 Dec;11(6):533-42. doi: 10.1007/s11892-011-0223-x. PMID 21912932
- [Background] Knip M, Veijola R, Virtanen SM, Hyoty H, Vaarala O, Akerblom HK. Environmental triggers and determinants of type 1 diabetes. Diabetes. 2005 Dec;54 Suppl 2:S125-36. doi: 10.2337/diabetes.54.suppl_2.s125. PMID 16306330
- [Background] Knip M, Simell O. Environmental triggers of type 1 diabetes. Cold Spring Harb Perspect Med. 2012 Jul;2(7):a007690. doi: 10.1101/cshperspect.a007690. PMID 22762021
- [Background] D'Angeli MA, Merzon E, Valbuena LF, Tirschwell D, Paris CA, Mueller BA. Environmental factors associated with childhood-onset type 1 diabetes mellitus: an exploration of the hygiene and overload hypotheses. Arch Pediatr Adolesc Med. 2010 Aug;164(8):732-8. doi: 10.1001/archpediatrics.2010.115. PMID 20679164
- [Background] Pociot F, Lernmark A. Genetic risk factors for type 1 diabetes. Lancet. 2016 Jun 4;387(10035):2331-2339. doi: 10.1016/S0140-6736(16)30582-7. PMID 27302272
- [Background] Rewers M, Ludvigsson J. Environmental risk factors for type 1 diabetes. Lancet. 2016 Jun 4;387(10035):2340-2348. doi: 10.1016/S0140-6736(16)30507-4. PMID 27302273
- [Background] Rubio-Cabezas O, Ellard S. Diabetes mellitus in neonates and infants: genetic heterogeneity, clinical approach to diagnosis, and therapeutic options. Horm Res Paediatr. 2013;80(3):137-46. doi: 10.1159/000354219. Epub 2013 Sep 18. PMID 24051999
- [Background] Soltesz G, Patterson CC, Dahlquist G; EURODIAB Study Group. Worldwide childhood type 1 diabetes incidence--what can we learn from epidemiology? Pediatr Diabetes. 2007 Oct;8 Suppl 6:6-14. doi: 10.1111/j.1399-5448.2007.00280.x. PMID 17727380